CLINICAL TRIAL: NCT01464736
Title: Impact of Aerobic Physical Training Associated With Noninvasive Ventilation on COPD Patient Functionality - A Controlled Randomized Study
Brief Title: Noninvasive Ventilation on Chronic Obstructive Pulmonary Disease (COPD) Patient Functionality
Acronym: kmarrara
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Kamilla Tays Marrara, Doutoranda em Fisioterapia pela Universidade Federal de São Carlos - UFSCar., Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFSCar
Record Dates: First submitted 2011-10-27; First posted 2011-11-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: aerobic exercise; noninvasive ventilation; functionality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Training Group (Experimental): This group performed aerobic physical training in treadmill.
  Interventions: Other: physical training
- NIV Trained (Experimental): This group performed aerobic physical training associated with ventilation in the bilevel modality (BiPAP®), using a nasal mask as an interface.
  On evaluation day, the levels of inspiratory positive airway pressure (IPAP) (between 10 and 15cmH2O) and expiratory positive airway pressure (EPAP) (between 4 and 6cmH2O) were defined, varying according to the comfort level of each patient.
  Interventions: Other: physical training

INTERVENTIONS:
Other: physical training — For both groups, the approximately hour-long sessions occurred three times a week on alternate days for six consecutive weeks (18 sessions). Each session began with five minutes of stretching that included the cervical muscles and the upper and lower limbs, which was followed by five minutes of warm-up on a treadmill at 2Km/h and 30 minutes of aerobic physical training at a constant 3% incline.
  Other Names: TFG: physical training group; PTGNIV: exercise plus bilevel ventilation group

SUMMARY:
On the following tests, there would be a greater increase in the functionality of COPD patients who underwent combined therapy than in those who only exercised: a set of activities of daily living (ADLs), the six-minute walk test (6MWT), an incremental symptom-limited cardiopulmonary test (CPT), and the physical functioning scale of the Short-Form 36 quality of life questionnaire (SF-36).

DETAILED DESCRIPTION:
Impact of aerobic exercise plus noninvasive ventilation (NIV) on the functionality of patients with COPD. Thirty patients (70.5 - 8.5 years) with COPD (forced expiratory volume in the first second 48.5 - 15.4% of predicted) were randomized into either a physical training group involving aerobic treadmill exercise (PTG, n=12) or an exercise plus bilevel ventilation group (PTGNIV, n=11) with sessions three times a week for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis
* with a forced expiratory volume in the first second (FEV1)/forced vital capacity (FVC)<70%
* clinical stability in the previous two months (i.e., no exacerbation of the disease).

Exclusion Criteria:

* decompensated heart failure or rheumatic, orthopedic or neuromuscular diseases that prevented the subjects from performing the tests due to exercise limitations;
* participation in a regular physical exercise program at the beginning of the study;
* noncompletion of one of the tests or the established protocol for any reason.

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-01; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Impact of aerobic exercise, either associated or not with NIV, by two positive pressure levels on COPD patient functionality. | 6 weeks
  It was measured by means of step-climbing repetitions and distance covered in the six-minute walk test as well as the CPT.

SECONDARY OUTCOMES:
Change in oxygen consumption. | 6 weeks
  It was evaluated through a MedGraphics VO2000 metabolic system which was operated via computer with Aerograph software and store the signals with the 20-second method at the peak of each activity in the set of ADLs and in the peak of CPT.
Change in metabolic rate. | 6 weeks.
  It was evaluated through a MedGraphics VO2000 metabolic system which was operated via computer with Aerograph software and store the signals with the 20-second method at the peak of each activity in the set of ADLs and in the peak of CPT.
Change in oxygenation. | 6 weeks.
  It was evaluated through a Dixtal® wrist oxymeter at the peak of each activity in the set of ADLs and in the peak of CPT.
Change in sensation of dyspnea. | 6 weeks
  It was evaluated through a modified Borg scale at the peak of each activity in the set of ADLs and in the peak of CPT.
Change in quality of life. | 6 weeks.
  It was evaluated through the SF-36 (domains: physical functioning, role-physical, and vitality).

CONTACTS AND LOCATIONS:
Overall Officials: Kamilla T Marrara, Doutoranda, Principal Investigator — Universidade Federal de São Carlos - UFSCar.; Diego M Marino, Doutorando, Study Chair — Universidade Federal de São Carlos - UFSCar.; Maurício Jamami, Professor, Study Chair — Universidade Federal de São Carlos - UFSCar.; Antônio D Oliveira Junior, Médico, Study Chair — Santa Casa de Misericórdia de São Carlos; Valéria A Pires Di Lorenzo, Professora, Study Director — Universidade Federal de São Carlos - UFSCar.
Locations (1):
- Universidade Federal de São Carlos - UFSCar., São Carlos, São Paulo, Brazil

REFERENCES:
- [Result] Casaburi R, Porszasz J, Burns MR, Carithers ER, Chang RS, Cooper CB. Physiologic benefits of exercise training in rehabilitation of patients with severe chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1997 May;155(5):1541-51. doi: 10.1164/ajrccm.155.5.9154855.
- [Result] Costes F, Agresti A, Court-Fortune I, Roche F, Vergnon JM, Barthelemy JC. Noninvasive ventilation during exercise training improves exercise tolerance in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2003 Jul-Aug;23(4):307-13. doi: 10.1097/00008483-200307000-00008. PMID 12894005
- [Result] Maltais F, Simard AA, Simard C, Jobin J, Desgagnes P, LeBlanc P. Oxidative capacity of the skeletal muscle and lactic acid kinetics during exercise in normal subjects and in patients with COPD. Am J Respir Crit Care Med. 1996 Jan;153(1):288-93. doi: 10.1164/ajrccm.153.1.8542131.
- [Result] Ambrosino N, Strambi S. New strategies to improve exercise tolerance in chronic obstructive pulmonary disease. Eur Respir J. 2004 Aug;24(2):313-22. doi: 10.1183/09031936.04.00002904. PMID 15332404
- [Result] Toledo A, Borghi-Silva A, Sampaio LM, Ribeiro KP, Baldissera V, Costa D. The impact of noninvasive ventilation during the physical training in patients with moderate-to-severe chronic obstructive pulmonary disease (COPD). Clinics (Sao Paulo). 2007 Apr;62(2):113-20. doi: 10.1590/s1807-59322007000200004. PMID 17505694
- [Result] Zuwallack R. Physical activity in patients with COPD: the role of pulmonary rehabilitation. Pneumonol Alergol Pol. 2009;77(1):72-6. No abstract available. PMID 19308913
- [Result] van 't Hul A, Gosselink R, Hollander P, Postmus P, Kwakkel G. Training with inspiratory pressure support in patients with severe COPD. Eur Respir J. 2006 Jan;27(1):65-72. doi: 10.1183/09031936.06.00036505. PMID 16387937
- [Result] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Result] Puhan MA, Mador MJ, Held U, Goldstein R, Guyatt GH, Schunemann HJ. Interpretation of treatment changes in 6-minute walk distance in patients with COPD. Eur Respir J. 2008 Sep;32(3):637-43. doi: 10.1183/09031936.00140507. Epub 2008 Jun 11. PMID 18550610
- [Result] Marrara KT, Marino DM, de Held PA, de Oliveira Junior AD, Jamami M, Di Lorenzo VA. Different physical therapy interventions on daily physical activities in chronic obstructive pulmonary disease. Respir Med. 2008 Apr;102(4):505-11. doi: 10.1016/j.rmed.2007.12.004. Epub 2008 Feb 1. PMID 18242069
- [Result] Brochard L, Mancebo J, Wysocki M, Lofaso F, Conti G, Rauss A, Simonneau G, Benito S, Gasparetto A, Lemaire F, et al. Noninvasive ventilation for acute exacerbations of chronic obstructive pulmonary disease. N Engl J Med. 1995 Sep 28;333(13):817-22. doi: 10.1056/NEJM199509283331301. PMID 7651472
- [Result] Brochard L. Non-invasive ventilation for acute exacerbations of COPD: a new standard of care. Thorax. 2000 Oct;55(10):817-8. doi: 10.1136/thorax.55.10.817. No abstract available. PMID 10992531